CLINICAL TRIAL: NCT03205059
Title: An Evidence-based Approach for Bullying Prevention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Health Promotion Associates, Inc. (Industry)
Responsible Party: Principal Investigator, Christopher Williams, Senior Vice President, National Health Promotion Associates, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R44HD074319-02 (NIH)
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Bullying; Cyberbullying; Substance Use; Substance Abuse
MeSH Terms: conditions — Bullying; Cyberbullying; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LST MS curriculum+ Bullying/Cyberbullying serious game (Experimental)
  Interventions: Behavioral: LST MS curriculum+ Bullying/Cyberbulling serious game
- LST MS curriculum (Active Comparator)
  Interventions: Behavioral: LST MS curriculum

INTERVENTIONS:
Behavioral: LST MS curriculum+ Bullying/Cyberbulling serious game — The prevention materials for middle school bullying and cyberbullying will (1) utilize both interactive classroom sessions and serious/educational games (digital games used to educate in an entertaining format); (2) positively change social norms surrounding bullying and cyberbulling; (3) challenge positive expectancies about bullying and cyberbullying; (4) enhance protective factors by building social, self-regulation, and relationship skills throughout the interactive learning and behavioral rehearsal; and (5) include booster sessions.
  Arms: LST MS curriculum+ Bullying/Cyberbullying serious game
Behavioral: LST MS curriculum — The evidence-based LifeSkills Training program has been successfully used as a universal, school-based substance abuse and violence prevention program for middle school youth. The goals of the LST program are to teach youth the personal self-management skills, social skills, and other life skills needed to successfully resist drug and alcohol use, navigate developmental tasks, increase resilience, and facilitate healthy psychosocial development.
  Arms: LST MS curriculum

SUMMARY:
This Phase II SBIR project is designed to address the critical public health problem of bullying and cyberbullying among middle school age youth. The project involves developing and testing bullying and cyberbullying prevention materials, including interactive classroom sessions and corresponding serious games, based on the evidence-based substance abuse prevention approach called Life Skills Training. The product has the potential to fill a gap in the intervention tools currently available to schools that can be widely disseminated throughout the country using existing marketing and dissemination channels and decrease the adverse consequences of bullying and cyberbullying as well as substance abuse.

ELIGIBILITY:
Inclusion Criteria:

* Middle school aged-youth

Exclusion Criteria:

* Significant cognitive impairment or severe learning disabilities, as screened by field staff at participating sites

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3000 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Change in bullying/cyberbullying perpetration in the past two years | Post-test (within 2 weeks of completing final session/module of the intervention), 12-month follow-up, 24-month follow-up
  The investigators will assess (via questionnaire) key study variables regarding bullying and cyberbullying and hypothesized risk and protective factors. These outcomes will be examined and compared in both the intervention group and the active comparator group at a post-test assessment and 12-month and 24-month follow-up assessments.

CONTACTS AND LOCATIONS:
Locations (1):
- National Health Promotion Associates, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: No